CLINICAL TRIAL: NCT02687139
Title: Study of PSMA-targeted 18F-DCFPyL PET/CT in the Evaluation of Patients With Renal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00075596
Record Dates: First submitted 2016-02-11; First posted 2016-02-22 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-DCFPyL PET/CT (Experimental)
  Interventions: Drug: 18F-DCFPyL; Procedure: PET/CT

INTERVENTIONS:
Drug: 18F-DCFPyL
Procedure: PET/CT — Positron Emission Tomography - Computed Tomography (PET/CT)

SUMMARY:
In this study the investigators aim to evaluate diagnostic utility of prostate-specific membrane antigen (PSMA)-targeted 18F-DCFPyL PET/CT in patients with renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed or histologically proven stage II-IV renal cell carcinoma
* Completed staging evaluation with computed tomography (CT) or magnetic resonance imaging (MRI) of the chest, abdomen and pelvis ≤90 days prior to study enrollment

Exclusion Criteria:

* History of other malignancy diagnosed within the last 3 years (with the exception of low risk prostate cancer, ductal carcinoma in situ of the breast, squamous cell carcinoma or basal cell carcinoma of the skin)
* Administered a radioisotope within 5 physical half-lives prior to study enrollment
* Pregnancy ((as determined in accordance with the policies of the positron emission tomography (PET) center))
* Intention to enroll in a blinded therapeutic clinical trial following Positron emission tomography-computed tomography (PET/CT)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Allaf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Meyer AR, Carducci MA, Denmeade SR, Markowski MC, Pomper MG, Pierorazio PM, Allaf ME, Rowe SP, Gorin MA. Improved identification of patients with oligometastatic clear cell renal cell carcinoma with PSMA-targeted 18F-DCFPyL PET/CT. Ann Nucl Med. 2019 Aug;33(8):617-623. doi: 10.1007/s12149-019-01371-8. Epub 2019 May 30. PMID 31147927

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-DCFPyL PET/CT: 18F-DCFPyL PET/CT: Positron Emission Tomography - Computed Tomography (PET/CT)
Period: Overall Study
Arm/Group | 18F-DCFPyL PET/CT
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 18F-DCFPyL PET/CT: Men and women of all races and ethnic groups are eligible for this study were encouraged to participate.
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 25
Age, Continuous [Median (Full Range); unit: years] | 60 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 18F-DCFPyL PET/CT Detected Sites of Metastatic Renal Cell Carcinoma (RCC)
Description: This was assessed to compare the sites of disease images of patients with RCC on conventional imaging with the images on the 18F-DCFPyL PET/CT to evaluate the sensitivity of DCFPyL PET/CT scans in detecting sites of disease compared to conventional imaging.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 34
Participants | 34

2. Primary Outcome: Number of Participants With a Correlation Between Radiotracer Uptake on 18F-DCFPyL PET/CT and Conventional Imaging
Description: This was assessed to Correlate Sites of Radiotracer Uptake on 18F-DCFPyL PET/CT With Conventional Imaging Findings.
Time Frame: 12 Months
Population: Only the first 14 participants enrolled in this study were assessed for this outcome and published at the time.
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 14
Participants | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 18F-DCFPyL PET/CT
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 3/34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-DCFPyL PET/CT (N=34)
Headache (Nervous system disorders) | 2 (2) — Headache post study injection
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT02687139/Prot_SAP_000.pdf